CLINICAL TRIAL: NCT04122989
Title: Validation of a Shared Decision-Making Tool, MS-SUPPORT, to Improve Decisions About Disease Modifying Therapies (DMT) for Multiple Sclerosis
Brief Title: Validation of a Shared Decision-Making Tool for Multiple Sclerosis
Acronym: MS-SUPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shared Decision Making Resources (Other)
Collaborators: EMD Serono (Industry); Multiple Sclerosis Association of America (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MS700568_0052
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial, with 1:1 randomization
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS-SUPPORT (Experimental): Group receives access to an online shared decision making tool (an interactive decision aid) for multiple sclerosis.
  Interventions: Other: MS-SUPPORT
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: MS-SUPPORT — MS-SUPPORT is a shared decision making tool designed to be used by patients and providers.
  Arms: MS-SUPPORT

SUMMARY:
This study evaluates a novel shared decision making tool for multiple sclerosis (MS). Half the patients will be given access to MS-SUPPORT before their scheduled appointment with their healthcare provider, the other half will not be given access.

DETAILED DESCRIPTION:
MS-SUPPORT is a novel shared-decision making tool. More specifically, it is a web-based decision aid (DA) that includes 'values clarification exercises' to support people with MS (PwMS) incorporate their preferences and values when faced with a DMT treatment decision. Each 'values clarification exercise' includes a written passage about a specific topic, with a series of questions. It covers topical domains related to living with MS and treatment decision making, including but not limited to lifestyle, tolerability, safety, risk tolerance, health goals, and personal values.

This validation study will evaluate the effect of using MS-SUPPORT on starting or switching DMTs, patient-provider communication, DMT adherence, Quality of Life (QoL), decision quality (the concordance of the treatment chosen, which includes no treatment, with the patient's values), quality of care, and decisional conflict. Participants will include adult patients with relapsing forms of MS and their MS healthcare providers (HCP). Patients will be randomized into one of two groups: MS-SUPPORT (intervention) or Usual Care (control).

ELIGIBILITY:
For MS patients:

Inclusion criteria:

* Able to read and write in English
* Live within the United States and receive MS care in the USA
* 18 years or older
* Having a diagnosis of a relapsing form of MS, including Relapsing Remitting Multiple Sclerosis (RRMS), active secondary progressive MS, and Clinically Isolated Syndrome (CIS)
* Having access to the internet
* Having a valid email address
* Have a healthcare provider who is managing their MS
* Having an upcoming appointment with an MS healthcare provider to manage their MS within the next 12 weeks

Exclusion criteria:

• Unable or unwilling to give informed consent

For HCPs:

Inclusion criteria:

* English-speaking
* Any HCP who manages a participating patient's MS

Exclusion criteria:

• Unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Start/Switch DMT | Quarterly during the 12 month follow-up after the index HCP visit.
  Proportion of MS patients that switch or start a disease modifying therapy (DMT).

SECONDARY OUTCOMES:
Patient-provider communication | Measured once, up to 2 months after the index HCP visit.
  We will use COMRADE, a validated patient self-report scale that measures communication, decision-making effectiveness, satisfaction with healthcare provider communication, and confidence in the decision made.
Adherence to DMT | Quarterly, up to 12 month follow-up after the index HCP visit.
  We will measure self-reported adherence to DMTs by asking patients to report the number of doses they took in the past month (or relevant dosing interval for that DMT if dosing is less frequent than one month) and divide that by the number of expected doses during that dosing interval. This value ranges from 0.0 to 1.0, with 1.0 indicating perfect adherence.
Decision Quality | Quarterly, up to 12 month follow-up after the index HCP visit.
  We will assess the extent to which the treatment chosen is consistent with the patient values by asking a question such as "My treatment plan is helping me achieve my treatment goals" and "My treatment plan reflects what's important to me when I think about the pros and cons of treatment."
Quality of Life--Healthy Days Core Module | Quarterly, up to 12 month follow-up after the index HCP visit.
  We will use the 4-item Healthy Days Core Module from the Health-Related Quality of Life (HR-QOL-14). This module assesses self-rated general health, including the number of days that the person is limited in their usual mental and physical activities. This measure was originally drawn from the State-based Behavioral Risk Factor Surveillance System (BRFSS) which has been used since 1993.
CAHPS Quality of Care | Measured once, up to 2 months after the index HCP visit.
  The 4-item communication items from the Patient Experience Measures from the Consumer Assessment of Healthcare Providers and Systems (CAHPS) Health Plan Survey coupled with a global assessment of their HCP and a single item from the CAHPS® Clinician & Group Surveys, Patient-Centered Medical Home (PCMH4: Someone from provider's office talked with patient about specific health goals) will be assessed.
Decision Conflict | Measured twice. First measurement, up to 1 month after starting the study. Second measurement, up to 2 months after the index HCP visit.
  A 4-item validated short-form of the original decisional conflict scale (SURE) will be used. These 4 items ask yes/no questions; the scoring algorithm combines the total score (maximum 4, minimum 0). Any score under 4 is considered a positive for decisional conflict.

CONTACTS AND LOCATIONS:
Overall Officials: Nananda Col, MD, MPH, MPP, Principal Investigator — Shared Decision Making Resources
Locations (1):
- Shared Decision Making Resources, Georgetown, Maine, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share all Individual Participant Data (IPD) that underlie results in a publication, ensuring that such data are deidentified.
Time Frame: Upon publication and for 1 year thereafter
Access Criteria: Contact the PI

REFERENCES:
- [Background] Edwards A, Elwyn G, Hood K, Robling M, Atwell C, Holmes-Rovner M, Kinnersley P, Houston H, Russell I. The development of COMRADE--a patient-based outcome measure to evaluate the effectiveness of risk communication and treatment decision making in consultations. Patient Educ Couns. 2003 Jul;50(3):311-22. doi: 10.1016/s0738-3991(03)00055-7. PMID 12900105
- [Background] Moriarty DG, Zack MM, Kobau R. The Centers for Disease Control and Prevention's Healthy Days Measures - population tracking of perceived physical and mental health over time. Health Qual Life Outcomes. 2003 Sep 2;1:37. doi: 10.1186/1477-7525-1-37. PMID 14498988
- [Background] Sepucha KR, Borkhoff CM, Lally J, Levin CA, Matlock DD, Ng CJ, Ropka ME, Stacey D, Joseph-Williams N, Wills CE, Thomson R. Establishing the effectiveness of patient decision aids: key constructs and measurement instruments. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S12. doi: 10.1186/1472-6947-13-S2-S12. Epub 2013 Nov 29. PMID 24625035
- [Background] Elwyn G, O'Connor A, Stacey D, Volk R, Edwards A, Coulter A, Thomson R, Barratt A, Barry M, Bernstein S, Butow P, Clarke A, Entwistle V, Feldman-Stewart D, Holmes-Rovner M, Llewellyn-Thomas H, Moumjid N, Mulley A, Ruland C, Sepucha K, Sykes A, Whelan T; International Patient Decision Aids Standards (IPDAS) Collaboration. Developing a quality criteria framework for patient decision aids: online international Delphi consensus process. BMJ. 2006 Aug 26;333(7565):417. doi: 10.1136/bmj.38926.629329.AE. Epub 2006 Aug 14. PMID 16908462
- [Background] Pieterse AH, de Vries M, Kunneman M, Stiggelbout AM, Feldman-Stewart D. Theory-informed design of values clarification methods: a cognitive psychological perspective on patient health-related decision making. Soc Sci Med. 2013 Jan;77:156-63. doi: 10.1016/j.socscimed.2012.11.020. Epub 2012 Nov 27. PMID 23219164
- [Background] Reynolds MW, Stephen R, Seaman C, Rajagopalan K. Persistence and adherence to disease modifying drugs among patients with multiple sclerosis. Curr Med Res Opin. 2010 Mar;26(3):663-74. doi: 10.1185/03007990903554257. PMID 20070144
- [Result] Col NF, Solomon AJ, Springmann V, Garbin CP, Ionete C, Pbert L, Alvarez E, Tierman B, Hopson A, Kutz C, Berrios Morales I, Griffin C, Phillips G, Ngo LH. Whose Preferences Matter? A Patient-Centered Approach for Eliciting Treatment Goals. Med Decis Making. 2018 Jan;38(1):44-55. doi: 10.1177/0272989X17724434. Epub 2017 Aug 14. PMID 28806143
- [Result] Col NF, Solomon AJ, Springmann V, Ionete C, Alvarez E, Tierman B, Kutz C, Morales IB, Griffin C, Ngo LH, Jones DE, Phillips G, Hopson A, Pbert L. Evaluation of a Novel Preference Assessment Tool for Patients with Multiple Sclerosis. Int J MS Care. 2018 Nov-Dec;20(6):260-267. doi: 10.7224/1537-2073.2017-021. PMID 30568563